CLINICAL TRIAL: NCT03729830
Title: Prospective Evaluation of Open Irrigated Ablation Catheters With High Resolution Mapping to Treat Paroxysmal Atrial Fibrillation
Acronym: INTERRUPT AF
Status: Completed | Type: Observational
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Other Study IDs: 92249986
Record Dates: First submitted 2018-11-01; First posted 2018-11-05 (Actual); Results first posted 2026-01-21 (Actual); Last update posted 2026-01-21 (Actual); Status verified 2025-12

CONDITIONS: Paroxysmal Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

INTERVENTIONS:
Device: Boston Scientific Open Irrigated Ablation Catheters — The BSC Open-Irrigated catheters are designed to deliver RF energy to catheter tip electrode for cardiac ablation. The BSC OI catheters incorporate an open-irrigated cooling mechanism through a tip that is partitioned into two chambers. The proximal chamber circulates normal saline (0.9 %) within the tip to cool the proximal electrode and mitigate overheating while the distal chamber allows the fluid to flow through six irrigation holes into the patient's vasculature, thereby cooling the tip/tissue interface.

SUMMARY:
To obtain data for the Rhythmia™ Mapping System in conjunction with Boston Scientific Open-Irrigated (OI) Catheters for ablation of Paroxysmal Atrial Fibrillation (PAF) according to current international and local guidelines.

Primary objective: To assess acute and long-term outcomes for the Rhythmia Mapping System in conjunction with Boston Scientific Open-Irrigated Ablation Catheters to treat de novo Paroxysmal Atrial Fibrillation. De Novo PAF is defined as subjects undergoing first ablation procedure for PAF with no prior left atrial ablation (RF, Cryo, Surgical).

DETAILED DESCRIPTION:
STUDY OBJECTIVE(S) -- To obtain data for the Rhythmia™ Mapping System in conjunction with Boston Scientific Open-Irrigated (OI) Catheters for ablation of Paroxysmal Atrial Fibrillation (PAF) according to current international and local guidelines.

PRIMARY OBJECTIVE -- To assess acute and long-term outcomes for the Rhythmia Mapping System in conjunction with Boston Scientific Open-Irrigated Ablation Catheters to treat de novo Paroxysmal Atrial Fibrillation. De Novo PAF is defined as subjects undergoing first ablation procedure for PAF with no prior left atrial ablation (RF, Cryo, Surgical).

INDICATION(S) FOR USE -- Study devices will be used per approved Indications for Use for each geography.

DEVICES / SYSTEM USED IN THE STUDY -- The study will include the following Boston Scientific Open-Irrigated Catheters in geographies where commercially approved for PAF ablation:

* Blazer Open-Irrigated Ablation Catheter
* IntellaNav Open-Irrigated Ablation Catheter
* IntellaNav MiFi Open-Irrigated Ablation Catheter
* IntellaTip MiFi Open-Irrigated Ablation Catheter
* Rhythmia Mapping System Gen 1or Rhythmia HDx, equipped with Software 1.4 or any successive commercially approved versions.
* IntellaMap Orion Catheter

CONTROL DEVICE -- There are no control devices in this study

STUDY DESIGN -- Prospective, non-randomized, multicenter (global), post approval clinical study (PAS). All subjects fitting the enrollment criteria, signing the consent and undergoing the index procedure with the study devices will be followed up for three years to complete the PAS design mandated from the FDA to collect post-market data for Boston Scientific Open-Irrigated Catheters and will be followed for three years.

PLANNED NUMBER OF SUBJECTS -- The study will enroll 415 subjects.

PLANNED NUMBER OF SITES / COUNTRIES -- The study is global (US, EU, Asia-Pacific) with 25-50 centers. A minimum of 50% of the sites will be selected from the US. No study site will be allowed to contribute more than 41 subjects (10% of the 415 enrollments requirement).

FOLLOW-UP SCHEDULE -- Study Follow-ups are at: pre-discharge, 1 month (phone check), 3 months (blanking period), 6 months (phone check), 12 months, 24 months and 36 months.

STUDY DURATION -- Study is expected to be completed in approximately five years (12-24 month enrollment period with three year follow-up).

PARTICIPANT DURATION -- The study duration for each subject is expected to be approximately three years.

ELIGIBILITY:
Inclusion Criteria:

1. History of recurrent symptomatic Paroxysmal Atrial Fibrillation, defined as AFib that terminates spontaneously or with intervention within seven days of onset. Minimum documentation includes a physician's note indicating recurrent self-terminating Atrial Fibrillation AND one electrocardiographically documented AF episode within 6 months prior to enrollment.
2. Subjects who are eligible for an ablation procedure for Paroxysmal Atrial Fibrillation with the Rhythmia Mapping system according to current international and local guidelines
3. Subjects who are eligible for an ablation procedure for Paroxysmal Atrial Fibrillation with a Boston Scientific Open-Irrigated Ablation Catheter according to current international and local guidelines
4. Subjects who are willing and capable of providing informed consent
5. Subjects who are willing and capable of participating in all testing associated with this clinical investigation at an approved clinical investigational center
6. Subjects whose age is 20 years or above, or who are of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

1. Subjects enrolled in any other concurrent clinical study, with the exception of local mandatory governmental registries and observational studies/registries, without the written approval from Boston Scientific
2. Subjects unable or unwilling to complete follow-up visits and examination for the duration of the study
3. Subjects who have undergone any previous left atrial cardiac ablation (RF, Cryo, surgical)
4. Subjects who have undergone any cardiac ablation within 30 days prior to enrollment
5. Unrecovered/unresolved Adverse Events from any previous invasive procedure
6. Life expectancy <= three years per physician opinion
7. Women of childbearing potential who are, or plan to become, pregnant during the time of the study (method of assessment upon physician's discretion)
8. Known cardiac thrombus within 60 days prior to enrollment
9. History of CVA, TIA or PE within 90 days prior to enrollment
10. Implanted pacemaker, ICD, or CRT leads within 90 days prior to enrollment
11. Implanted Left atrial appendage closure device prior to the index procedure
12. Prosthetic mitral or tricuspid heart valves (subjects with successful mitral valve repair allowed- annular ring constitutes repair)
13. Left atrial diameter greater than 5.5cm
14. Documented or suspected stenosis of any pulmonary veins.
15. Atrial fibrillation secondary to electrolyte imbalance, thyroid disease, or reversible or non-cardiac cause.
16. Contraindication for anticoagulation
17. Clinically significant mitral valve regurgitation or stenosis per investigator discretion.
18. Any cardiac surgery ≤ 90 days from consent date.
19. Any electrocardiographically documented episode of Persistent AFib, defined as AFib lasting longer than 7 days from onset.

Min Age: 20 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Subjects included in the INTERRUPT AF study should be selected from the investigator's general patient population indicated for catheter ablation of PAF.
Sampling Method: Non-Probability Sample
Enrollment: 415 (Actual)
Dates: Start 2019-03-04 (Actual); Primary Completion 2024-05-03 (Actual); Study Completion 2024-05-03 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Oussama Wazni, Principal Investigator — The Cleveland Clinic
Locations (26):
- United States (18):
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Torrance Memorial Medical Center, Torrance, California
  - Broward General Medical Center, Miami, Florida
  - AdventHealth Orlando, Orlando, Florida
  - St. Lukes Idaho Cardiology Associates, Boise, Idaho
  - University of Chicago Hospital, Chicago, Illinois
  - St. John's Hospital, Springfield, Illinois
  - University of Iowa Hospitals and Clinics, Iowa City, Iowa
  - Nebraska Heart Institute, Lincoln, Nebraska
  - Dartmouth Hitchcock Medical Center, Lebanon, New Hampshire
  - Catholic Medical Center, Manchester, New Hampshire
  - Kaleida Health, Buffalo, New York
  - Bethesda North Hospital, Cincinnati, Ohio
  - Cleveland Clinic Foundation, Cleveland, Ohio
  - Lehigh Valley Hospital, Allentown, Pennsylvania
  - HeartPlace Mid-Cities EP, Bedford, Texas
  - Orion Medical, Pasadena, Texas
  - Christus Trinity Mother Frances Health System, Tyler, Texas
- Germany (2):
  - Staedtisches Klinikum Karlsruhe, Karlsruhe
  - Juedisches Krankenhaus Berlin, Mitte
- Japan (2):
  - Kokura Memorial Hospital, Fukuoka-ken
  - Yokosuka Kyosai Hospital, Kanagawa Prefecture
- Centre Hospitalier Princesse Grace, Monaco, Monaco
- South Korea (2):
  - Keimyung University Dongsan Medical Center, Daegu
  - Korea University Medical Center, Seoul
- Papworth Hospital, Cambridge, United Kingdom

IPD SHARING:
Plan to Share IPD: No
No requests for study data have been made at this time, however Boston's Scientific's policy on data sharing can be found at http://www.bostonscientific.com/en-US/data-sharing-requests.html

RESULTS

PARTICIPANT FLOW:
Groups:
- INTERRUPT AF Clinical Study: Patients who underwent treatment with a Boston Scientific open-irrigated ablation catheter for the treatment of paroxysmal atrial fibrillation in conjunction with the Rhymthia Mapping System
  Devices/Systems used in the study:
  Boston Scientific Open-Irrigated Catheters:
  * IntellaNav Open-Irrigated Ablation Catheter
  * IntellaNav MiFi Open-Irrigated Ablation Catheter
  * IntellaTip MiFi Open-Irrigated Ablation Catheter
  * Rhythmia Mapping System Gen 1or Rhythmia HDx, equipped with Software 1.4 or any successive commercially approved versions.
  * IntellaMap Orion Catheter
Period: Overall Study
Arm/Group | INTERRUPT AF Clinical Study
Started | 415 (Consented subjects= 415 * Treated = 383 * Intent= 32 Subjects who were enrolled in the study but did not undergo ablation procedure within 60 days from consent signature date)
Procedure | 383
Completed | 148
Not Completed | 267
Not completed — Active at study close | 136
Not completed — Subject withdrew consent | 40
Not completed — Intent | 32
Not completed — Lost to Follow-up | 31
Not completed — research facility closed down | 9
Not completed — Death | 5
Not completed — Physician Decision | 4
Not completed — No longer meets protocol criteria | 3
Not completed — Protocol Violation | 6
Not completed — Sponsor withdrew subject | 1

BASELINE CHARACTERISTICS:
Arm/Group | INTERRUPT AF Clinical Study
Number analyzed (Participants) | 415
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: 414 analyzed instead of 415 as 1 patient withdrew from the study prior to providing this information
  years
    number analyzed (Participants) | 414
    (all) | 63.2 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: 414 analyzed instead of 415 as 1 patient withdrew from the study prior to providing this information
  Participants
    number analyzed (Participants) | 414
    Female | 155
    Male | 259
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Population: Race not reported for 8 subjects
  Participants
    Race: number analyzed (Participants) | 407
    Race: White | 282
    Race: Black | 10
    Race: Hispanic or Latino | 5
    Race: Asian | 95
    Race: Race Not Disclosed | 15
Region of Enrollment [Number; unit: participants]
  South Korea | 21
  Monaco | 6
  United States | 278
  Japan | 82
  United Kingdom | 4
  Germany | 24
Weight [Mean (Standard Deviation); unit: kg] — Population: Weight not reported for 2 subjects
  kg
    number analyzed (Participants) | 413
    (all) | 87.7 (24.2)
Height [Mean (Standard Deviation); unit: cm] — Population: Height not reported for 2subjects
  cm
    number analyzed (Participants) | 413
    (all) | 172.1 (10.2)
BMI [Mean (Standard Deviation); unit: kg/m^2] — Population: BMI not reported for 2 subjects
  kg/m^2
    number analyzed (Participants) | 413
    (all) | 29.4 (7.2)
Resting Systolic BP [Mean (Standard Deviation); unit: mmHG] — Population: Resting systolic BP not reported for 3 subjects
  mmHG
    number analyzed (Participants) | 412
    (all) | 132.6 (19.6)
Resting Diastolic BP [Mean (Standard Deviation); unit: mmHG] — Population: Resting diastolic BP not reported for 3 subjects
  mmHG
    number analyzed (Participants) | 412
    (all) | 78.4 (12.6)
Resting Heart Rate [Mean (Standard Deviation); unit: bpm] — Population: Resting heart rate not reported for 3 subjects
  bpm
    number analyzed (Participants) | 412
    (all) | 68.4 (15.1)
Cardiac Non-Arrhythmic [Count of Participants; unit: Participants] — Participants can be counted more than once in the appropriate category.
  Participants
    Cardiovascular Disease | 227
    Cardiomyopathy | 34
    Valvular Disease | 21
    Coronary Artery Disease | 74
    Cardiac Disease Other | 15
    Congestive Heart Failure | 25
    Cerebrovascular Disease | 4
    Peripheral Vascular Disease | 12
    Hypertension | 159
    Pulmonary Hypertension | 5
    Hyperlipidemia | 119
    Coagulopathy - Hypercoagulable State - Clotting Disorder | 11
    Transient Ischemic Attack (TIA) CVA or PE | 19
    Cardiac thrombus | 5
    Other cardiovascular disease occurred | 194
    No history of cardiac disease | 186
Cardiac Procedure History [Count of Participants; unit: Participants] — Population: 414 analyzed instead of 415 as 1 patient withdrew from the study prior to providing this information
  Participants
    number analyzed (Participants) | 414
    Cardiac procedures | 77
    Cardiac ablations | 28
    None | 309
Noncardiac Comorbidities [Count of Participants; unit: Participants] — Participants can be counted more than once in the appropriate category.
  Participants
    COPD | 24
    Diabetes | 60
    Hepatic Disease | 7
    Neurological Disease | 11
    Renal Disease | 17
    GI Bleeding | 12
    Sleep Disordered Breathing | 76
    Other comorbidities | 97
    Non-study hospitalization | 16
    None | 211
Arrhythmia History [Count of Participants; unit: Participants] — Participants can be counted more than once in the appropriate category. Population: Arrhythmia history not reported for 3 patients
  Participants
    Ventricular Arrhythmia Occurred: number analyzed (Participants) | 412
    Ventricular Arrhythmia Occurred | 56
    No Ventricular Arrhythmias: number analyzed (Participants) | 412
    No Ventricular Arrhythmias | 357
    Atrial Arrhythmia Occurred: number analyzed (Participants) | 412
    Atrial Arrhythmia Occurred | 412
    No Atrial Arrhythmias: number analyzed (Participants) | 412
    No Atrial Arrhythmias | 1
    ORT or AVRT: number analyzed (Participants) | 412
    ORT or AVRT | 5
    Focal Atrial Tachycardia: number analyzed (Participants) | 412
    Focal Atrial Tachycardia | 2
    Accessory Pathway: number analyzed (Participants) | 412
    Accessory Pathway | 9
    Paroxysmal Atrial Fibrillation: number analyzed (Participants) | 412
    Paroxysmal Atrial Fibrillation | 412
    Atrial Tachycardia: number analyzed (Participants) | 412
    Atrial Tachycardia | 25
    Atrial Flutter: number analyzed (Participants) | 412
    Atrial Flutter | 103
    Atrial Arrhythmia Other: number analyzed (Participants) | 412
    Atrial Arrhythmia Other | 16
    Brady Arrhythmia Occurred: number analyzed (Participants) | 412
    Brady Arrhythmia Occurred | 108
    Sinus Bradycardia: number analyzed (Participants) | 412
    Sinus Bradycardia | 92
    Sinus Node Dysfunction: number analyzed (Participants) | 412
    Sinus Node Dysfunction | 11
    Sick Sinus Syndrome Chronotropic Incompetence: number analyzed (Participants) | 412
    Sick Sinus Syndrome Chronotropic Incompetence | 10
    Sinus arrest: number analyzed (Participants) | 412
    Sinus arrest | 2
    AV Block 1: number analyzed (Participants) | 412
    AV Block 1 | 23
    AV Block 2: number analyzed (Participants) | 412
    AV Block 2 | 1
    Brady Arrhythmia Other: number analyzed (Participants) | 412
    Brady Arrhythmia Other | 2

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants Safety Event-free at 12 Months Post Procedure
Description: This measure reports the observed safety event -free rate at 12 Months follow up. The safety events are a composite of acute primary safety events (events occurring within seven days post-procedure or hospital discharge, whichever is later), and chronic primary safety events (events occurring through 3- or 12-months post-procedure, as listed below).
  Acute primary safety endpoint events are defined as the following:
  * Death
  * Myocardial infarction (MI)
  * Vagal Nerve Injury/Gastroparesis
  * Transient ischemic attack (TIA)
  * Stroke/Cerebrovascular accident (CVA)
  * Thromboembolism
  * Pericarditis
  * Cardiac tamponade/perforation
  * Pneumothorax
  * Vascular access complications
  * Pulmonary edema/heart failure
  * AV block
  Chronic primary safety endpoint events are defined as the following occurring through:
  3 Months post-procedure 12 Months post-procedure
  * Atrial esophageal fistula
  * Pericardial effusion
  * Pulmonary vein stenosis (symptomatic and requiring intervention)
Time Frame: 12 months
Population: This analysis includes all treatment and attempt subjects, including those with missing data.
Measure: Number; unit: Number of Participants
Groups:
- Treatment With Ablation Catheter: Patients who undergo treatment with a Boston Scientific open-irrigated ablation catheter for the treatment of paroxysmal atrial fibrillation in conjunction with the Rhymthia Mapping System
  Treatment with Blazer Open-Irrigated Ablation Catheter, IntellaNav Open-Irrigated Ablation Catheter, IntellaNav MiFi Open-Irrigated Ablation Catheter, or IntellaTip MiFi Open-Irrigated Ablation Catheter: Patients will be treated with an ablation catheter
Arm/Group | Treatment With Ablation Catheter
Number analyzed (Participants) | 383
Number of Participants | 368

2. Primary Outcome: Number of Participants Effectiveness Event -Free at 12 Months Post Procedure
Description: The primary effectiveness endpoint is defined as the event-free rate at 12 months post-procedure.
  Primary effectiveness events are defined as:
  * Acute procedural failure
  * More than one repeat procedure during the blanking period (90 days post index procedure)
  * Documented atrial fibrillation, or new onset of atrial flutter or atrial tachycardia event (≥ 30 seconds in duration from an event monitor or Holter, or from a 10 second 12-lead EKG) between 91 days and 365 days post index procedure
  * Any of the following interventions for atrial fibrillation, or new onset of atrial flutter or atrial tachycardia between 91 days and 365 days post index procedure:
  * Repeat procedure
  * Cardioversion
  * Prescribed any AAD*
    * AADs for endpoint will consist of all Class I/III and any Class II/IV medications taken for control of AF/AT/AFL recurrence
Time Frame: 12 Months
Measure: Number; unit: Number of Participants
Arm/Group | Treatment With Ablation Catheter
Number analyzed (Participants) | 383
Number of Participants | 218

3. Secondary Outcome: Number of Participants Event Free Rate (Secondary)
Description: The secondary effectiveness endpoint is defined as the event-free at 12 months post-procedure.
  Secondary effectiveness events are defined as:
  * Acute procedural failure
  * More than one repeat procedure during the blanking period (90 days post index procedure)
  * Documented symptomatic atrial fibrillation, or new onset of atrial flutter or atrial tachycardia event (≥ 30 seconds in duration from an event monitor or Holter, or from a 10 second 12-lead EKG) between 91 days and 365 days post index procedure
  * Any of the following interventions for atrial fibrillation, or new onset of atrial flutter or atrial tachycardia between 91 days and 365 days post index procedure:
  * Repeat procedure
  * Cardioversion
  * Prescribed a higher dose of any AAD* documented at baseline
  * Prescribed a new AAD* not documented at baseline
    * AADs for endpoint will consist of all Class I/III and any Class II/IV medications taken for control of AF/AT/AFL recurrence
Time Frame: 12 Months
Measure: Count of Participants; unit: Participants
Arm/Group | Treatment With Ablation Catheter
Number analyzed (Participants) | 383
Participants | 102

ADVERSE EVENTS:
Time Frame: 12 months
Description: There is only one arm in the study- Treatment Arm (383 subjects). Intent subjects (32) are not considered a study arm Consented subjects= 415
  * Treated = 383
  * Intent= 32 Subjects who were enrolled in the study but did not undergo ablation procedure within 60 days from consent signature date
Arm/Group | Treatment With Ablation Catheter
All-Cause Mortality (participants affected / at risk) | 5/383
Serious Adverse Events (participants affected / at risk) | 135/383
Other Adverse Events (participants affected / at risk) | 46/383
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Ablation Catheter (N=383)
Procedure related general adverse reaction (Surgical and medical procedures) | 1 (1)
Angina/Chest pain (Surgical and medical procedures) | 7 (7)
Hematological (Blood and lymphatic system disorders) | 1 (1)
Aortic stenosis (Cardiac disorders) | 2 (2)
Atrial Fibrillation (Cardiac disorders) | 46 (54)
Atrial Flutter (Cardiac disorders) | 12 (13)
Atrial Flutter, not specified (Cardiac disorders) | 1 (2)
Atrial Tachycardia/Other SVT (eg AVRT, AVNRT, EAT) (Cardiac disorders) | 3 (3)
Atrial tachycardia (Cardiac disorders) | 1 (1)
Atypical (Type II) Atrial Flutter (Cardiac disorders) | 4 (4)
Cardiac arrest (Cardiac disorders) | 1 (1)
Dyspnea - Heart failure (Cardiac disorders) | 2 (2)
Exacerbation of pre-existing condition (Cardiac disorders) | 1 (1)
Heart failure symptoms - Unspecified (Cardiac disorders) | 3 (3)
Mitral regurgitation (Cardiac disorders) | 1 (1)
Mitral stenosis (Cardiac disorders) | 1 (1)
Multiple heart failure symptoms (Cardiac disorders) | 3 (3)
Palpitations (Cardiac disorders) | 1 (1)
Peripheral edema - Heart failure (Cardiac disorders) | 1 (1)
Premature Ventricular Contractions (PVC) (Cardiac disorders) | 1 (1)
Sinus bradycardia (Cardiac disorders) | 3 (3)
Tachy-brady syndrome (Cardiac disorders) | 1 (1)
Tachyarrhythmia (Cardiac disorders) | 1 (1)
Ventricular Tachycardia (VT)/Monomorphic VT (Cardiac disorders) | 2 (2)
Endocrine (Endocrine disorders) | 3 (3)
Gastrointestinal (Gastrointestinal disorders) | 11 (13)
Abnormal laboratory values (General disorders) | 6 (6)
Adverse reaction - Medication (General disorders) | 2 (2)
Chest pain - Other (General disorders) | 6 (7)
Death (General disorders) | 1 (1)
Dizziness (General disorders) | 2 (2)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 3 (3)
Panniculectomy (General disorders) | 1 (1)
Physical trauma (General disorders) | 7 (7)
Syncope (General disorders) | 3 (3)
bleeding from hemodialysis site (General disorders) | 1 (1)
Infection - Unrelated (non study) procedure or device (Infections and infestations) | 1 (1)
Systemic infection (Infections and infestations) | 2 (2)
Adverse reaction - Abnormal labs - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Adverse reaction - Anesthesia/Sedation - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Adverse reaction - Hypertension - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Adverse reaction - Hypotension - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Adverse reaction - Neurological (non-TIA, non-stroke) - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Adverse reaction - Pulmonary - EP procedure (Injury, poisoning and procedural complications) | 3 (3)
Conduction pathway injury (pacemaker implantation) - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Exacerbation of existing condition - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Hematoma (Injury, poisoning and procedural complications) | 1 (1)
Major bleeding/hemorrhage requiring transfusion (Injury, poisoning and procedural complications) | 1 (1)
Myocardial perforation with tamponade (Injury, poisoning and procedural complications) | 3 (3)
Other - Unrelated (non study) procedure or device (ICD EOL) (Injury, poisoning and procedural complications) | 1 (1)
Other - Unrelated (non study) procedure or device (LV Lead revision) (Injury, poisoning and procedural complications) | 1 (1)
Other - Unrelated (non study) procedure or device (RV Lead revision) (Injury, poisoning and procedural complications) | 1 (1)
Pericardial effusion - EP procedure (Injury, poisoning and procedural complications) | 6 (6)
Pericarditis - EP procedure (Injury, poisoning and procedural complications) | 2 (2)
Pleural Effusion - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Post-surgical infection/sepsis - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Pseudoaneurysm - EP procedure (Injury, poisoning and procedural complications) | 2 (2)
Stroke (ischemic) - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Transient Ischemic Attack (TIA) - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 6 (7)
Cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 5 (5)
Neurological (Nervous system disorders) | 6 (6)
Elevated threshold - RA Lead (Product Issues) | 1 (1)
Oversensing - RV PG System (Product Issues) | 1 (1)
Genitourinary (Renal and urinary disorders) | 4 (4)
Renal (Renal and urinary disorders) | 3 (4)
Pulmonary (Respiratory, thoracic and mediastinal disorders) | 11 (17)
Adverse reaction - Hypotension (Vascular disorders) | 1 (1)
Cerebrovascular Accident (CVA) - unspecifed (Vascular disorders) | 2 (3)
Coronary Artery Disease (Vascular disorders) | 2 (2)
Distal thromboemboli (Vascular disorders) | 1 (1)
Edema (Vascular disorders) | 1 (1)
Hematoma - Unrelated (non study) procedure or device (Vascular disorders) | 2 (2)
Hypertension/Hypertensive Crisis (Vascular disorders) | 1 (1)
Hypotension/Orthostatic Hypotension (Vascular disorders) | 2 (2)
Myocardial infarction (Vascular disorders) | 6 (6)
Pseudoaneurysm with hematoma (Vascular disorders) | 1 (1)
Pulmonary Embolism (PE) (Vascular disorders) | 1 (1)
Transient Ischemic Attack (TIA) (Vascular disorders) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Treatment With Ablation Catheter (N=383)
Adverse reaction - General - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Angina/Chest pain - Post EP procedure (Injury, poisoning and procedural complications) | 8 (8)
Puncture site hematoma - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Vasospasm - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Atrial Fibrillation (AF) (Cardiac disorders) | 5 (6)
Atrial Flutter (Cardiac disorders) | 1 (1)
Atrial Flutter, not specified (Cardiac disorders) | 2 (2)
Sinus bradycardia (Cardiac disorders) | 1 (1)
Gastrointestinal (Gastrointestinal disorders) | 1 (1)
Head, eyes, ears, nose, throat (HEENT) (General disorders) | 1 (1)
Syncope (General disorders) | 1 (1)
Adverse reaction - Abnormal labs - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Adverse reaction - Anesthesia/Sedation - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Adverse reaction - Gastrointestinal - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Adverse reaction - Genitourinary/Renal - EP procedure (Injury, poisoning and procedural complications) | 2 (2)
Adverse reaction - Neurological (non-TIA, non-stroke) - EP procedure (Injury, poisoning and procedural complications) | 2 (2)
Angina/Chest pain - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Embolism - Air - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Exacerbation of existing condition - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Hematoma - EP procedure (Injury, poisoning and procedural complications) | 2 (2)
Inadvertent injury to adjacent structure - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Minor oozing/bleeding - EP procedure (Injury, poisoning and procedural complications) | 3 (3)
Pain (non-cardiovascular) - EP procedure (Injury, poisoning and procedural complications) | 5 (5)
Pericarditis - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Post-surgical wound discomfort - EP procedure (Injury, poisoning and procedural complications) | 6 (7)
Stroke (ischemic) - EP procedure (Injury, poisoning and procedural complications) | 1 (1)
Ablation-EP Related~Other (Injury, poisoning and procedural complications) | 3 (3)
Musculoskeletal (Musculoskeletal and connective tissue disorders) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2019-02-12): https://cdn.clinicaltrials.gov/large-docs/30/NCT03729830/Prot_000.pdf
  • Statistical Analysis Plan (2020-12-17): https://cdn.clinicaltrials.gov/large-docs/30/NCT03729830/SAP_001.pdf